CLINICAL TRIAL: NCT03604341
Title: Cannabinoid Analgesia for Medical Abortion: A Randomized Controlled Trial
Brief Title: Cannabinoids for Pain Control During Medical Abortion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Jeffrey Jensen, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OHSU IRB 18195
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Medical Abortion; Pain
Keywords: Medical Abortion; Pain; Cannabis
MeSH Terms: conditions — Pain; Marijuana Abuse | interventions — Dronabinol; Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gestational age up to 10w0d - Dronabinol (Experimental): Women with gestational age up to 10 weeks 0 days will be randomized to Dronabinol 5mg Cap or placebo
  Interventions: Drug: Dronabinol 5mg Cap
- Gestational age up to 10w0d - Placebo (Placebo Comparator): Women with gestational age up to 10 weeks 0 days will be randomized to Dronabinol 5mg Cap or placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dronabinol 5mg Cap — Subjects randomized to Dronabinol 5mg Cap and ibuprofen 800mg for pain
  Other Names: Dronabinol
  Arms: Gestational age up to 10w0d - Dronabinol
Other: Placebo — Subjects randomized to placebo and ibuprofen 800mg for pain
  Arms: Gestational age up to 10w0d - Placebo

SUMMARY:
The objective of this study is to determine if a synthetic cannabis derivative, dronabinol, in addition to ibuprofen, decreases maximum pain scores compared to ibuprofen and placebo in women undergoing medical abortion. Results of this study will help providers counsel patients regarding cannabis use during medical abortion.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled trial comparing pain levels in women undergoing medical abortion with one of two regimens: ibuprofen 800mg and a 5mg oral dronabinol versus ibuprofen 800mg and placebo given at the time of misoprostol administration. This study will include 62 women undergoing medical abortion. Women will be randomized to dronabinol 5mg oral versus placebo. The primary outcome will be maximum reported pain score within 24 hours of misoprostol administration.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years or older
* Consented for elective medical abortion
* Pregnancy with intrauterine gestational sac up to 10 0/7 weeks, dated by ultrasound
* Able and willing to receive text messages via phone
* English speaking
* Able and willing to give informed consent and agree to the study terms
* Have assistance at home; no motor vehicle use while taking study medications

Exclusion Criteria:

* Desires to continue pregnancy or currently breastfeeding
* Lack of access to cell phone and texting capabilities
* Prior participation in this study
* Early pregnancy failure
* Contraindications to the study medications: Marinol or marijuana derivatives, sesame oil, Ibuprofen
* Contraindications to medical abortion with Mifepristone or Misoprostol
* History of methadone, buprenorphine or heroin use within the last year
* History of a seizure disorder
* Used marijuana 5 or more days in the last week
* History of any adverse effects associated with prior use of recreational or medical marijuana products, or sensitivity/allergy to Marinol.

Ages: 21 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers or used for future research.

REFERENCES:
- [Derived] Colwill AC, Alton K, Bednarek PH, Bayer LL, Jensen JT, Garg B, Beardsworth K, Edelman A. Cannabinoids for Pain Control During Medical Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2020 Jun;135(6):1289-1295. doi: 10.1097/AOG.0000000000003850. PMID 32459420

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants failed to meet the inclusion criteria after enrollment and were not assigned to a treatment group.
Period: Overall Study
Arm/Group | Gestational Age up to 10w0d - Dronabinol | Gestational Age up to 10w0d - Placebo
Started | 35 | 35
Completed | 33 | 33
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gestational Age up to 10w0d - Dronabinol | Gestational Age up to 10w0d - Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (6.5) | 28.6 (5.0) | 28.3 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Non-Hispanic | 20 | 22 | 42
  Other | 15 | 13 | 28
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Maximum Self-reported Pain Score on a Numeric Rating Scale
Description: Women will text responds to surveys within 24 hours after misoprostol administration indicating their maximum self-reported pain using an 11-point numeric rating scale (NRS 0-10) where 0=no pain and 10=worst possible pain.
Time Frame: 24 hours after misoprostol administration
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Gestational Age up to 10w0d - Dronabinol | Gestational Age up to 10w0d - Placebo
Number analyzed (Participants) | 33 | 33
score on a scale | 7 [6 to 8] | 7 [5 to 8]

ADVERSE EVENTS:
Time Frame: from enrollment to 21 days after abortion procedure
Arm/Group | Gestational Age up to 10w0d - Dronabinol | Gestational Age up to 10w0d - Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 2/35 | 0/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gestational Age up to 10w0d - Dronabinol (N=35) | Gestational Age up to 10w0d - Placebo (N=35)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT03604341/Prot_SAP_000.pdf